CLINICAL TRIAL: NCT02855177
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Parallel-group Study To Assess The Safety, Tolerability, And Pharmacokinetics With 2-weeks Of Dosing Of Pf-06427878 In Overweight-obese, Otherwise Healthy Adult Subjects
Brief Title: A Multiple Dose Safety And Pharmacokinetic (PK) Study Of PF-06427878 In Overweight-Obese, Otherwise Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7871005
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
Keywords: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be administered as an extemporaneously prepared suspension every 8 hours for 14 days
  Interventions: Drug: Placebo
- PF-06427878 (Experimental): PF-06427878 will be administered as an extemporaneously prepared suspension every 8 hours for 14 days
  Interventions: Drug: PF-06427878

INTERVENTIONS:
Drug: Placebo — Placebo as suspension administered every 8 hours, with food
  Arms: Placebo
Drug: PF-06427878 — 500 mg suspension administered every 8 hours, with food
  Arms: PF-06427878

SUMMARY:
PF-06427878 is a new compound proposed for the treatment of hyperlipidemia. The primary purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics after 2 weeks of dosing of PF-06427878 in overweight-obese, otherwise healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential.
* Body Mass Index (BMI) of >=25 kg/m2; and a total body weight >50 kg
* Subjects with liver fat >=6% and <=20%

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary,gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Emergent Treatment-Related Adverse Events (AEs) | Day -2 to Day 44
Change from baseline in clinical laboratory tests | Day 1 to Day 22
Change from baseline in vital signs | Day 0 to Day 22
Change from baseline in cardiac conduction intervals assessed via 12-lead electrocardiogram | Day 0 to Day 22

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06427878 on day 1 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06427878 on day 1 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Area Under the Curve for PF-06427878 during the dosing interval (AUCtau) on day 1 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06427878 on day 14 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06427878 on day 14 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Area Under the Curve for PF-06427878 during the dosing interval (AUCtau) on day 14 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Plasma Decay Half-Life (t1/2) for PF-06427878 on day 14 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Apparent Volume of Distribution (Vz/F) of PF-06427878 on day 14 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Apparent Oral Clearance (CL/F) of PF-06427878 on day 14 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Minimum Observed Plasma Concentration (Cmin) for PF-06427878 on day 14 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Peak:Trough ratio of PF-06427878 on day 14 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Accumulation ratio for Area Under the Curve during the dosing interval (Rac(AUCtau)) for PF-06427878 on day 14 relative to day 1 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Accumulation ratio for Maximum Observed Plasma Concentration (Rac(Cmax)) for PF-06427878 on day 14 relative to day 1 | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post dose
Amount of PF-06427878 excreted in urine (Ae) on day 14 | 0-8 hours post dose
Percent of dose excreted in urine as PF-06427878 (Ae%) on day 14 | 0-8 hours post dose
Renal clearance of PF-06427878 (CLr) on day 14 | 0-8 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - California Clinical Trials Medical Group, Glendale, California
  - Qps-Mra, Llc, South Miami, Florida

REFERENCES:
- [Derived] Amin NB, Carvajal-Gonzalez S, Purkal J, Zhu T, Crowley C, Perez S, Chidsey K, Kim AM, Goodwin B. Targeting diacylglycerol acyltransferase 2 for the treatment of nonalcoholic steatohepatitis. Sci Transl Med. 2019 Nov 27;11(520):eaav9701. doi: 10.1126/scitranslmed.aav9701. PMID 31776293
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7871005&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo-controlled%2C+Parallel-group+Study+To+Assess+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+With+2-weeks+Of+Dosing+Of+Pf-06427878+In+Overweight-obese%2C+Otherwise+Healthy+Adult+Subjects